CLINICAL TRIAL: NCT01681121
Title: A Twelve-week, Double-blind, Placebo-controlled, Randomized, Parallel-group, Multi-center Study of the Safety and Efficacy of ADX-N05 in the Treatment of Excessive Daytime Sleepiness in Subjects With Narcolepsy
Brief Title: A Study of the Safety and Effectiveness of ADX-N05 for Excessive Daytime Sleepiness in Subjects With Narcolepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADX-N05 202
Record Dates: First submitted 2012-09-05; First posted 2012-09-07 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Narcolepsy
MeSH Terms: conditions — Narcolepsy | interventions — solriamfetol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADX-N05 (Experimental): ADX-N05 to be taken once a day for 12 weeks
  Interventions: Drug: ADX-N05
- Placebo (Placebo Comparator): Placebo to match ADX-N05 to be taken once a day for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ADX-N05 — 150 mg once a day for 4 weeks followed by 300 mg once a day for 8 weeks
  Arms: ADX-N05
Drug: Placebo — One capsule placebo to match ADX-N05 to be taken for 4 weeks followed by 2 capsules placebo to match ADX-N05 to be taken for 8 weeks
  Arms: Placebo

SUMMARY:
This is a study to evaluate the safety and effectiveness of ADX-N05 compared to placebo in the treatment of excessive daytime sleepiness in adults with narcolepsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of narcolepsy
* Good general health
* Willing and able to comply with the study design and schedule and other requirements

Exclusion Criteria:

* If female, pregnant or lactating
* Customary bedtime later than midnight
* History of significant medical condition, behavioral, or psychiatric disorder (including suicidal ideation), or surgical history
* Any other clinically relevant medical, behavioral or psychiatric disorder other than narcolepsy that is associated with excessive sleepiness
* History of significant cardiovascular disease
* Body mass index > 34
* Excessive caffeine use - > 600 mg/day of caffeine or > 6 cups of coffee/day
* History of alcohol or drug abuse within the past 2 years
* Nicotine dependence that has an effect on sleep

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ward, MD, Study Director — Aerial BioPharma, LLC
Locations (28):
- United States (28):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Pulmonary Associates, Phoenix, Arizona
  - Stanford Sleep Medicine Center, Redwood City, California
  - Pacific Research Network, San Diego, California
  - Sleep-Alertness Disorders Center, Aurora, Colorado
  - PAB Clinical Research, Brandon, Florida
  - Clinical Research Group of St. Petersburg, St. Petersburg, Florida
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - Sleep Disorders Center of Georgia, Atlanta, Georgia
  - SleepMed of Central Georgia, Macon, Georgia
  - Chicago Research Center, Chicago, Illinois
  - Community Research, Crestview Hills, Kentucky
  - Kentucky Research Group, Louisville, Kentucky
  - The Center for Sleep and Wake Disorders, Chevy Chase, Maryland
  - Pulmonary and Critical Care Associates of Baltimore, Towson, Maryland
  - Neurocare, Inc., Newton, Massachusetts
  - Minnesota Lung Center and Sleep Institute, Edina, Minnesota
  - Washington University, St Louis, Missouri
  - Rex Sleep Disorders Center, Raleigh, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Mercy St. Vincent Medical Center, Toledo, Ohio
  - Center for Sleep Medicine, Philadelphia, Pennsylvania
  - SleepMed of South Carolina, Columbia, South Carolina
  - Future Search Trials of Neurology, Austin, Texas
  - Sleep Medicine Associates of Texas, Dallas, Texas
  - Todd J. Swick, MD, PA, Houston, Texas
  - Metroplex Pulmonary and Sleep Center, McKinney, Texas
  - Sleep Therapy and Research Center, San Antonio, Texas

REFERENCES:
- [Derived] Ruoff C, Swick TJ, Doekel R, Emsellem HA, Feldman NT, Rosenberg R, Bream G, Khayrallah MA, Lu Y, Black J. Effect of Oral JZP-110 (ADX-N05) on Wakefulness and Sleepiness in Adults with Narcolepsy: A Phase 2b Study. Sleep. 2016 Jul 1;39(7):1379-87. doi: 10.5665/sleep.5968. PMID 27166238

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ADX-N05 | Placebo
Started | 44 | 49
Completed | 36 | 38
Not Completed | 8 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ADX-N05 | Placebo | Total
Number analyzed (Participants) | 44 | 49 | 93
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41 (12.33) | 36.7 (11.71) | 38.7 (12.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 14 | 19 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Average Sleep Latency Time (in Minutes) as Determined From the Maintenance of Wakefulness Test (MWT) for ADX-N05 300 mg vs. Placebo at Last Assessment.
Description: The MWT is a validated objective measure of the ability to stay awake for a defined period of time. The primary analysis was a comparison of treatments vs. control groups on change from Baseline to last available post-Baseline assessment (Week 12/Last Assessment) in the average sleep latency time (in minutes) averaged across the first four trials of the MWT using a two-sample t-test.
Time Frame: Baseline up to Week 12/Last Assessment post-dose.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ADX-N05 | Placebo
Number analyzed (Participants) | 40 | 45
minutes | 12.8 (10.28) | 2.1 (7.88)

2. Primary Outcome: Number of Participants With Improved Clinical Global Impression of Change (CGI-C) Scores for ADX-N05 vs. Placebo at Last Assessment
Description: The CGI-C scale rated the change in the participant's condition as compared to the Baseline visit on a 7-point scale ranging from a minimum of "Very much improved" to a maximum of "Very much worse." The proportion of subjects experiencing at least minimal improvement on the CGI-C was calculated and summarized for each of the treatment groups at Week 4 and the last available post-Baseline assessment (Week 12/Last Assessment). The CGI-C scale consists of the following ratings: 1-Very Much improved, 2-Much improved, 3-Minimally improved, 4-No change, 5-Minimally worse, 6-Much worse, 7-Very much worse; a rating of 1 indicates a better outcome, and a rating of 7 indicates a worse outcome. Improvement was defined as a CGI-rating of 1, 2, or 3.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | ADX-N05 | Placebo
Number analyzed (Participants) | 43 | 47
Participants | 37 | 18

3. Secondary Outcome: Change From Baseline in the Average Sleep Latency Time (in Minutes) as Determined From the Maintenance of Wakefulness Test (MWT) (Average of the First Four Trials) Following Four Weeks of Treatment With ADX-N05 150 mg vs. Placebo
Description: The MWT is a validated objective measure of the ability to stay awake for a defined period of time. The MWT consisted of five 40-minute trials separated by 2 hour intervals.
  This secondary analysis repeated the primary analysis for effects at the end of Week 4.
Time Frame: Baseline up to Week 4 post-dose.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ADX-N05 | Placebo
Number analyzed (Participants) | 40 | 45
minutes | 9.5 (8.38) | 1.4 (7.59)

4. Secondary Outcome: Change From Baseline in Sleep Latency Time (in Minutes) as Determined From Each of the 5 Individual MWT Trials for ADX-N05 vs. Placebo at Week 4
Description: The MWT is a validated objective measure of the ability to stay awake for a defined period of time. The MWT consisted of five 40-minute trials separated by 2 hour intervals.
  This secondary analysis repeated the primary analysis for effects for the five MWT trials analyzed separately at Week 4.
Time Frame: Baseline up to Week 4 post-dose.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ADX-N05 | Placebo
Number analyzed (Participants) | 40 | 45
minutes
  Trial 1 | 11.7 (12.50) | 1.6 (9.86)
  Trial 2 | 9.7 (12.51) | 1.0 (9.01)
  Trial 3 | 9.9 (11.44) | 1.3 (9.86)
  Trial 4 | 6.8 (10.56) | 1.8 (7.64)
  Trial 5 | 5.4 (9.10) | -4.0 (12.28)

5. Secondary Outcome: Change From Baseline in Sleep Latency Time (in Minutes) as Determined From Each of the 5 Individual MWT Trials for ADX-N05 vs. Placebo at Last Assessment
Description: The MWT is a validated objective measure of the ability to stay awake for a defined period of time. The MWT consisted of five 40-minute trials separated by 2 hour intervals.
  This secondary analysis repeated the primary analysis for effects for the five MWT trials analyzed separately at the last available post-Baseline assessment (Week 12/Last Assessment).
Time Frame: Baseline up to Week 12/Last Assessment post-dose.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ADX-N05 | Placebo
Number analyzed (Participants) | 40 | 45
minutes
  Trial 1 | 15.5 (13.84) | 2.6 (10.65)
  Trial 2 | 13.4 (15.31) | 2.7 (10.97)
  Trial 3 | 11.4 (12.62) | 2.0 (10.83)
  Trial 4 | 10.8 (13.85) | 1.0 (6.92)
  Trial 5 | 8.2 (12.73) | -1.6 (13.12)

6. Secondary Outcome: Change From Baseline in Epworth Sleepiness Scale (ESS) Scores for ADX-N05 vs. Placebo at Week 4
Description: The ESS is a questionnaire intended to measure daytime sleepiness. In this test, participants answer questions with regard to the level of sleepiness they experienced over approximately the 7 days prior to the assessment while performing eight common, non-stimulating activities. The ESS total score range is 1 to 24. Each activity is rated on a 4-point scale ranging from a minimum of "would never doze" to a maximum of "a high chance of dozing." Thus, the ESS scale range is as follows: 0=would never doze, 1=slight chance of dozing, 2=moderate chance of dozing, 3=high chance of dozing; 0 indicates a better outcome, and 3 indicates a worse outcome. A negative mean change value indicates a decrease in score from baseline and an improvement in daytime sleepiness.
Time Frame: Baseline up to Week 4 post-dose.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ADX-N05 | Placebo
Number analyzed (Participants) | 40 | 45
score on a scale | -5.6 (5.28) | -2.4 (4.60)

7. Secondary Outcome: Change From Baseline in ESS Scores for ADX-N05 vs. Placebo at Last Assessment
Description: as for outcome 6
Time Frame: Baseline up to Week 12/Last Assessment post-dose.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ADX-N05 | Placebo
Number analyzed (Participants) | 43 | 47
score on a scale | -8.5 (5.75) | -2.5 (5.13)

8. Secondary Outcome: Number of Participants With Improved Clinical Global Impression of Change (CGI-C) Scores for ADX-N05 vs. Placebo at Week 4
Description: as for outcome 2
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | ADX-N05 | Placebo
Number analyzed (Participants) | 40 | 45
Participants | 32 | 23

9. Secondary Outcome: Number of Participants With Improved Patient Global Impression Change (PGI-C) Scores for ADX-N05 vs. Placebo at Week 4
Description: The Patient Global Impression - Change (PGI-C) scale was completed by the subject at the Weeks 1, 2, 4, 6, 8, and 12 visits. The CGI-C scale rated the change in the participant's condition as compared to the Baseline visit on a 7-point scale ranging from a minimum of "Very much improved" to a maximum of "Very much worse." The proportion of subjects experiencing at least minimal improvement on the CGI-C was calculated and summarized for each of the treatment groups at Week 4 and the last available post-Baseline assessment (Week 12/Last Assessment). The CGI-C scale consists of the following ratings: 1-Very Much improved, 2-Much improved, 3-Minimally improved, 4-No change, 5-Minimally worse, 6-Much worse, 7-Very much worse; a rating of 1 indicates a better outcome, and a rating of 7 indicates a worse outcome. Improvement was defined as a CGI-rating of 1, 2, or 3.
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | ADX-N05 | Placebo
Number analyzed (Participants) | 40 | 45
Participants | 33 | 20

10. Secondary Outcome: Number of Participants With Improved PGI-C Scores for ADX-N05 vs. Placebo at Last Assessment
Description: as for outcome 9
Time Frame: Week 12/Last Assessment
Measure: Count of Participants; unit: Participants
Arm/Group | ADX-N05 | Placebo
Number analyzed (Participants) | 43 | 47
Participants | 40 | 18

ADVERSE EVENTS:
Arm/Group | ADX-N05 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/49
Serious Adverse Events (participants affected / at risk) | 2/44 | 0/49
Other Adverse Events (participants affected / at risk) | 21/44 | 12/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADX-N05 (N=44) | Placebo (N=49)
Conversion Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ADX-N05 (N=44) | Placebo (N=49)
Headache (Nervous system disorders) | 7 | 5
Insomnia (Nervous system disorders) | 6 | 1
Dizziness (Nervous system disorders) | 3 | 1
Initial Insomnia (Nervous system disorders) | 2 | 2
Middle Insomnia (Nervous system disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 6 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 3
Upper Respirstory Tract Infection (Infections and infestations) | 2 | 4
Nasophanyngitis (Infections and infestations) | 2 | 1
Anxiety (Psychiatric disorders) | 5 | 0
Agitation (Psychiatric disorders) | 3 | 0
Bruxism (Psychiatric disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other